CLINICAL TRIAL: NCT05086471
Title: Performance Evaluation of the NaviCam SB Capsule Endoscope System in Comparison to the PillCam SB3 Capsule System for the Diagnosis of Small Bowel Diseases
Brief Title: Performance Evaluation of the NaviCam SB Capsule Endoscope System for the Diagnosis of Small Bowel Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Changhai Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NaviCam SB
Record Dates: First submitted 2021-09-30; First posted 2021-10-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2021-10

CONDITIONS: Small Bowel Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NaviCam SB (Experimental): After gastrointestinal preparation, the enrolled patients swallow NaviCam SB and the PillCam SB3 capsules approximately 40 minutes apart in a randomized order for small bowel capsule endoscopy.
  Interventions: Device: NaviCam SB
- PillCam SB3 (Other): After gastrointestinal preparation, the enrolled patients swallow NaviCam SB and the PillCam SB3 capsules approximately 40 minutes apart in a randomized order for small bowel capsule endoscopy.
  Interventions: Device: PillCam SB3

INTERVENTIONS:
Device: NaviCam SB — Subjects swallow two types of SB capsules approximately 40 minutes apart in a randomized order. During the capsule endoscopy, the doctor can view the small bowel images taken by the capsules in real time.
  Arms: NaviCam SB
Device: PillCam SB3 — Subjects swallow two types of SB capsules approximately 40 minutes apart in a randomized order. During the capsule endoscopy, the doctor can view the small bowel images taken by the capsules in real time.
  Arms: PillCam SB3

SUMMARY:
This study uses a comparative method to evaluate the performance of the NaviCam SB capsule endoscope system in comparison to the PillCam SB3 capsule system for the diagnosis of small bowel diseases.

DETAILED DESCRIPTION:
This study adopts a prospective and self-controlled design. The subjects are adult patients (≥18 years old) who have symptoms of small bowel disease or suspected GI bleeding; Subjects swallow two types of SB capsules approximately 40 minutes apart in a randomized order. During the capsule endoscopy, the doctor can view the small bowel images taken by the capsules in real time. This study adopts a method of independent image reading in the participating centers. Two physicians of digestive endoscopy respectively review the images captured by the experimental capsule and the control capsule for normal versus abnormal findings, type of findings and categorization (lesions, polyps, bleeding, etc.), capsule transit time, reading time, and image quality.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old) who have symptoms of small bowel disease or suspected GI bleeding;
2. Those need capsule endoscopy because the recurring GI symptoms cannot be explained by other imaging methods;
3. Those can understand and accept this study protocol and voluntarily sign an informed consent.

Exclusion Criteria:

1. Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule;
2. Patient with known gastrointestinal motility disorders;
3. Patient with known or suspected gastrointestinal obstruction, stenosis or fistula;
4. Patient with known or suspected delayed gastric emptying;
5. Patient suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions;
6. Patient has any allergy or other known contraindication or intolerance to the medications used in the study;
7. Patient has any condition, which precludes compliance with study and/or device instructions;
8. Women who are either pregnant or nursing at the time of screening;
9. Concurrent participation in another clinical trial using any investigational drug or device;
10. Patient suffers from a life-threatening condition;
11. Patients with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters;
12. Patients with pace-maker or implantable cardioverter other implantable electronic medical device;
13. Patient with an easily magnetized metal part;
14. Patient requires endoscopic placement of the capsule;
15. Others considered by the investigator not suitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic agreement rate | 14 days
  The diagnosis of subjects by the two types of small bowel capsule endoscopes through independent image reading, that is, the agreement between the two systems with respect to the diagnosis of normal or abnormal subject.

SECONDARY OUTCOMES:
Intestinal transit time | 14 days
  The time from capsule swallowing to capsule excretion
Ease of swallowing the capsule | 14 days
  The subject's supervisor determines how easy it is to swallow the capsule and which of the following feelings is very easy, easy, moderate, difficult, or very difficult.
diagnosis rate | 14 days
  Comparison of the diagnosis rate (examination results within one week before or after enrollment) with other standard mucosal imaging tools (upper GI endoscopy, enteroscopy, colonoscopy, etc.)
Quality of small bowel images | 14 days
  Comparison of the quality of small intestine pictures taken with the two capsules
Image reading time | 14 days
  Comparison of the reading times of the two capsules

CONTACTS AND LOCATIONS:
Overall Officials: XiaoHua Hou, MD.PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong Univerdity of Science and Technology; Rong Lin, MD.PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong Univerdity of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong Univerdity of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No